CLINICAL TRIAL: NCT01198704
Title: Study of Factors Predicting Tumor Recurrence After Liver Transplantation for Hepatocellular Carcinoma
Brief Title: Study of Factors Predicting Tumor Recurrence After Liver Transplantation for Hepatocellular Carcinoma (HCC)
Acronym: EFAPRE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: AOM07237
Record Dates: First submitted 2010-04-29; First posted 2010-09-10 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Hepatocellular Carcinoma; Liver Cirrhosis; Evidence of Liver Transplantation
Keywords: Hepatocellular carcinoma; Cirrhosis; Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and serum sample (28 ml at M0, M3, M6) Tissues (one pretransplant, hepatic explant, potential resection)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCC patients: Patients notified on the national waiting list for hepatic transplant
  Interventions: Other: search of factors predicting tumor recurrence

INTERVENTIONS:
Other: search of factors predicting tumor recurrence — Morphological, chronological, anatomy-pathological and molecular search

SUMMARY:
Results of liver transplantation, the best theoretical treatment for HCC, are limited by tumor recurrence. In order to limit this risk Milan criteria was proposed in 1996. However, these criteria are to restrictive and approximately 40% of patients denied by Milan criteria may be cured by liver transplantation.

The purpose of this study was thus to prospectively evaluate factors predicting tumor recurrence after liver transplantation for HCC and then to reassess criteria for liver transplantation.

DETAILED DESCRIPTION:
In this study, the investigators studied the predictive value of imaging techniques such as CT, MRI, PET scan, of serological markers and molecular markers assessed before liver transplantation at listing.

The investigators also evaluated the predictive value of tumor growing during the waiting time (imaging and serological).

Finally, the investigators compared pre-LT data and explanted liver analysis to evaluate accuracy of liver biopsy and of imaging.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* Hepatocellular carcinoma diagnosed by AASLD criteria or liver biopsy
* Listing for Liver transplantation for HCC fulfilling or not Milan criteria
* No extra-hepatic spread
* No vascular involvement

Exclusion Criteria:

* Salvage transplantation
* Transplantation contra-indication
* Evaluation for Liver transplantation older than 1 month
* Incidental HCC

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient notified on the waiting list for hepatic transplant
Sampling Method: Non-Probability Sample
Enrollment: 372 (Actual)
Dates: Start 2009-01; Primary Completion 2017-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Predictive factors of HCC recurrence | at 2 years after Liver transplantation for HCC (modified by amendment on 17/10/2013)

SECONDARY OUTCOMES:
Predictive factors of tumor-free recurrence | at 3 years
Predictive factors of overall survival at 5 years | at 5 years
Predictive factors of drop-out | during the waiting time
Radio-pathological correlation | end of the study
Correlation of HCC differentiation between liver biopsy and explant liver | at 32 month

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Decaens, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Clinique Universitaire d'Hépato-gastroentérologie, Grenoble, France